CLINICAL TRIAL: NCT00116064
Title: A Randomised Trial to Compare the Efficacy and Safety of Intranasal Lorazepam and Intramuscular Paraldehyde in the Treatment of Convulsions in Children
Brief Title: Intranasal Lorazepam Versus Intramuscular Paraldehyde in Paediatric Convulsions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kamuzu University of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03/04/248
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2006-07-21 (Estimated); Status verified 2005-06

CONDITIONS: Status Epilepticus; Convulsions
Keywords: intranasal; lorazepam; paediatric; convulsions
MeSH Terms: conditions — Status Epilepticus; Seizures

INTERVENTIONS:
Drug: intranasal lorazepam
Drug: intramuscular paraldehyde

SUMMARY:
The purpose of this study is to evaluate intranasal lorazepam in paediatric status epilepticus. This is a potentially, more effective, safer and cheaper treatment for a common paediatric medical emergency compared to our present first line therapy intramuscular paraldehyde.

DETAILED DESCRIPTION:
The ideal first line anticonvulsant agent would be one that can be safely and easily given at a primary health care facility. It should be quick acting, have minimal cardiorespiratory side effects and have a relatively prolonged effect and be cheap. No combination of drug or delivery system fully satisfies these criteria. There are no large published studies evaluating intranasal lorazepam in paediatric status epilepticus. Given its favourable pharmacokinetics and potential practical advantages, we wished to assess the efficacy and safety of intranasal delivery of lorazepam compared to intramuscular paraldehyde, our existing first line anticonvulsant agent in the treatment of acute seizures in children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 2 months and 12 years
* Presenting with generalised convulsions

Exclusion Criteria:

* Any child who had received an anticonvulsant agent within 1 hour of presentation
* Seizure stopped with rapid cooling or treatment of hypoglycaemia
* Features consistent with organophosphate poisoning, hepatic or hypertensive encephalopathy

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 156
Dates: Start 2004-07; Study Completion 2005-06

PRIMARY OUTCOMES:
whether the presenting seizure stopped or not with a single dose of assigned anticonvulsant agent within 10 minutes of administration

SECONDARY OUTCOMES:
time from drug administration to cessation of convulsion
frequency of episodes requiring 2 or more anticonvulsant agents
continuous blood pressure and oxygen saturation for 30 minutes post drug administration
seizure recurrence within 24 hours of cessation of presenting convulsion
survival/death

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Molyneux, MRCPCH FFAEM, Study Director — Kamuzu University of Health Sciences; Shafique Ahmad, MRCPCH FFAEM, Principal Investigator — Kamuzu University of Health Sciences
Locations (1):
- Paediatric Emergency Department, Queen Elizabeth Central Hospital, Blantyre, Malawi

REFERENCES:
- [Result] Ahmad S, Ellis JC, Kamwendo H, Molyneux E. Efficacy and safety of intranasal lorazepam versus intramuscular paraldehyde for protracted convulsions in children: an open randomised trial. Lancet. 2006 May 13;367(9522):1591-7. doi: 10.1016/S0140-6736(06)68696-0. PMID 16698412